CLINICAL TRIAL: NCT04193293
Title: A Phase 1b/2 Study of Duvelisib in Combination With Pembrolizumab in Subjects With Recurrent or Metastatic Head and Neck Squamous Cell Cancer
Brief Title: A Study of Duvelisib in Combination With Pembrolizumab in Head and Neck Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to low enrollment.
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-0145-130
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma of the Head and Neck; Head and Neck Cancer; PI3K-δ,γ; PI3K Inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — duvelisib; pembrolizumab; Immune Checkpoint Inhibitors; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Duvelisib + Pembrolizumab (Experimental): Stage 1: Duvelisib twice daily (BID) for 1 week followed by combination therapy with duvelisib BID + pembrolizumab every 3 weeks (q3w) (Cycle 1 was 4 weeks consisting of the 1-week duvelisib monotherapy lead-in period followed by 1 dose of pembrolizumab in combination with 3 additional weeks of continuous dosing of duvelisib; subsequent cycles were 3 weeks).
  Stage 2: Duvelisib BID + pembrolizumab q3w in 3-week cycles.
  Interventions: Drug: Duvelisib; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Duvelisib — Phosphoinositide 3-kinase (PI3K) Inhibitor
  Other Names: VS-0145; Copiktra
Biological: Pembrolizumab — Immunotherapy (programmed cell death protein 1 [PD-1] inhibitor)
  Other Names: PD-1 inhibitor; anti-PD-1; Keytruda

SUMMARY:
This study was designed to assess the safety and preliminary efficacy of duvelisib in combination with pembrolizumab in participants with recurrent or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
This was a non-randomized, open-label Phase 1b/2 study designed to evaluate safety, tolerability, and preliminary efficacy of duvelisib in combination with pembrolizumab in participants with R/M HNSCC who were eligible for pembrolizumab monotherapy based on the current pembrolizumab prescribing information.

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group performance status ≤ 1
* Histologically or cytologically confirmed diagnosis of recurrent or metastatic head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx that was considered incurable by local therapies
* Eligible for pembrolizumab monotherapy based on the current prescribing information for pembrolizumab (Keytruda 2019)
* Must have had 0 to 2 prior therapies for R/M HNSCC
* At least 1 measurable lesion (which has not been previously irradiated) according to Response Evaluation Criteria in Solid Tumors version 1.1
* For stage 1 only: Must have had at least 1 other lesion that could be biopsied and willing to undergo a pretreatment and on-treatment biopsy of the available tumor lesion
* For stage 1 only: Must have been willing to undergo a pretreatment and on-treatment biopsy of the available tumor lesion
* Adequate organ function defined by the following laboratory parameters:

  * Absolute neutrophil count ≥ 1.5 × 10^9/liter (L)
  * Platelet count ≥ 100 × 10^9/L
  * Hemoglobin level ≥ 9.0 grams/deciliter (dL)
  * A serum creatinine level < 1.5 milligrams/dL, or
  * Estimated creatinine clearance value ≥ 60 milliliters/minute (as determined by the Cockcroft-Gault method) for participants with creatinine levels > 1.5 × institutional upper limit of normal (ULN)
  * Total bilirubin level ≤ 1.5 × ULN (exception: participants with Gilbert's Syndrome may have a bilirubin level > 1.5 × ULN)
  * Aspartate aminotransaminase/serum glutamic-oxaloacetic transaminase and alanine aminotransferase/serum pyruvic transaminase levels ≤ 2.5 × ULN or ≤ 5 × ULN in participants with liver metastases
* International normalized ratio or prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, unless participant was receiving anticoagulant therapy in which case PT or aPTT must have been within therapeutic range of intended use of anticoagulants

Exclusion Criteria

* Previously treated with 3 or more systemic regimens given for recurrent and/or metastatic disease
* Received anticancer treatment, major surgery, or any investigational drug within 30 days or 5 half-lives, whichever is shorter, before the start of study intervention
* Received radiation therapy within 14 days before the start of study intervention, including, in addition (if necessary), the timeframe for resolution of any actual or anticipated toxicities from such radiation; Palliative radiation is allowed if > 7 days and any toxicity is ≤ Grade 1
* Previous treatment with a PI3K, PD-1 or programmed cell death ligand 1 inhibitor
* Have received organ or allogenic bone marrow or peripheral blood stem cell transplant
* History of drug-induced colitis or drug-induced pneumonitis; history or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function; tuberculosis treatment within 2 years prior to the start of study intervention; chronic liver disease or veno-occlusive disease/sinusoidal obstruction syndrome
* Active cytomegalovirus or Epstein-Barr virus infection; history of or known human immunodeficiency virus infection
* Ongoing treatment with chronic immunosuppressants or systemic steroids or treatment for systemic bacterial, fungal, or viral infection
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), or herpes zoster (VZV) at screening
* Concurrent administration of medications or foods that are strong inhibitors or inducers of cytochrome P450 3A. No prior use within 2 weeks before the start of study intervention Received a live or live attenuated vaccine within 6 weeks of first dose of duvelisib
* Unable to receive prophylactic treatment for pneumocystis, HSV, or VZV at screening
* Any active gastrointestinal dysfunction interfering with the participant's ability to be administered oral medications
* Known active central nervous system metastases and/or carcinomatous meningitis
* QT interval > 500 milliseconds (except for participants with a right or left bundle branch block)
* New York Heart Association Class III or IV congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated by the Sponsor due to low enrollment. Due to study termination and only 2 participants receiving treatment, there are concerns regarding participant confidentiality, therefore no data are being reported.
Period: Overall Study
Arm/Group | Duvelisib + Pembrolizumab
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated by the Sponsor. Due to study termination and only 2 participants receiving treatment, there are concerns regarding participant confidentiality, therefore no data are being reported.
Groups:
- Duvelisib + Pembrolizumab: Stage 1: Duvelisib BID for 1 week followed by combination therapy with duvelisib BID + pembrolizumab q3w (Cycle 1 was 4 weeks consisting of the 1-week duvelisib monotherapy lead-in period followed by 1 dose of pembrolizumab in combination with 3 additional weeks of continuous dosing of duvelisib; subsequent cycles were 3 weeks).
  Stage 2: Duvelisib BID + pembrolizumab q3w in 3-week cycles.
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Number of Participants With Dose-limiting Toxicities
Time Frame: 4 weeks or 28 days
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

2. Primary Outcome: Stage 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs as assessed by the Common Terminology Criteria for Adverse Events version 5 (CTCAE v5) as a measure of safety and tolerability of duvelisib in combination with pembrolizumab.
Time Frame: 6 months
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

3. Primary Outcome: Stage 1 and 2: Overall Response Rate (ORR)
Description: Proportion of participants achieving complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1).
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Stage 1: ORR
Description: Proportion of participants achieving complete CR or PR according to RECIST v 1.1.
Time Frame: Until documented progressive disease (PD), unacceptable toxicity, discontinuation criteria are met, withdrawal, or death (up to 2 years)
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Stage 1 and 2: Duration of Response (DOR)
Description: Time from response ≥ PR to documented disease progression according to RECIST v 1.1.
Time Frame: From first response until documented PD (up to 2 years)
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Stage 1 and 2: Progression-free Survival (PFS)
Description: Time from start of treatment to documented disease progression according to RECIST v 1.1, or death due to any cause.
Time Frame: From start of treatment until documented PD or death (up to 2.5 years)
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Stage 1 and 2: Overall Survival
Description: Time from start of treatment to death.
Time Frame: From start of treatment until death (up to 2.5 years)
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Stage 1 and 2: Maximum Observed Concentration [Cmax]
Description: Pharmacokinetics (PK) parameters for duvelisib (and metabolite IPI-656) determined using bioanalytical data and Population PK (POPPK) modeling.
Time Frame: Up to 5 cycles (46 weeks)
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Stage 1 and 2: Area Under the Curve [AUC]
Description: PK parameters for duvelisib (and metabolite IPI-656) determined using bioanalytical data and POPPK modeling.
Time Frame: Up to 5 cycles (46 weeks)
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Stage 1 and 2: Number of Participants With TEAEs
Description: Number of participants with TEAEs as assessed by CTCAE v5.0.
Time Frame: 24 months
Population: as for baseline characteristics
Arm/Group | Duvelisib + Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: This study was terminated by the Sponsor. Due to study termination and only 2 participants receiving treatment, there are concerns regarding participant confidentiality, therefore no data are being reported.
Description: This study was terminated by the Sponsor. Due to study termination and only 2 participants receiving treatment, there are concerns regarding participant confidentiality, therefore no data are being reported.
Arm/Group | Duvelisib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor due to low enrollment. Due to study termination and only 2 participants receiving treatment, there are concerns regarding participant confidentiality, therefore no data are being reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT04193293/Prot_SAP_000.pdf